CLINICAL TRIAL: NCT04753619
Title: Effectiveness of Niclosamide as Add-on Therapy to the Standard of Care Measures in COVID-19 Management (Randomized Controlled Clinical Trial)
Brief Title: Effectiveness of Niclosamide as Add-on Therapy to the Standard of Care Measures in COVID-19 Management
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Faiq Gorial, Professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO2021070003
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Covid-19; SARS Pneumonia
Keywords: Niclosamide; Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Niclosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Niclosamide group: NCS group (Experimental): NCL + standard therapy
  Interventions: Drug: Niclosamide Oral Tablet
- Control group (No Intervention): Control group

INTERVENTIONS:
Drug: Niclosamide Oral Tablet — * NCS 2 grams orally loading dose chewable then 1g every 8 hours in the first day, then on the 2nd day 1g x3 for 7 days. [ this means only in the first day 4 gm/d then on the second day 3g/d in 3 divided doses for 7 days]
  * If the participant requires mechanical ventilation over the course of the study, NGT may be administered via nasogastric (NG) or orogastric (OG) tube and, if possible, should be administered with a scheduled nasogastric (NG) or orogastric (OG) feeding.
  Other Names: Yomesan
  Arms: Niclosamide group: NCS group

SUMMARY:
Assessment of the Effectiveness of Niclosamide as Add on Therapy to the Standard of care Measures in COVID-19 Management in a randomized controlled clinical trial

DETAILED DESCRIPTION:
Protocol of therapy Niclosamaide Add on group

* NCS 2 grams orally loading dose chewable then 1g every 8 hours in the first day, then on the 2nd day 1g x3 for 7 days. [ this means only in the first day 4 gm/d then on the second day 3g/d in 3 divided doses for 7 days]
* If the participant requires mechanical ventilation over the course of the study, NGT may be administered via nasogastric (NG) or orogastric (OG) tube and, if possible, should be administered with a scheduled nasogastric (NG) or orogastric (OG) feeding.

Control group The patients in this group will receive only standard care which will include all or some of the following, according to the clinical condition of each patient:

* Acetaminophen 500mg on need
* Vitamin C 1000mg twice/ day
* Zinc 75-125 mg/day
* Vitamin D3 5000IU/day
* Azithromycin 250mg/day for 5 days
* Oxygen therapy/ C-Pap if needed
* Dexamethasone 6 mg/day or methylprednisolone 40mg twice per day, if needed
* Mechanical ventilation, if needed

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age above 18 years and of any gender.
2. Definite diagnosis of COVID-19 according to the WHO classification criteria ( 18).
3. Patients symptomatic for no more than three days for mild-moderate cases, no more than two days after being severe cases, and no more than one day after being critical cases.
4. Understands and agrees to comply with planned study procedures.

Exclusion Criteria:

1. Patients refuse to enrol in the study
2. Patients with hypersensitivity or severe adverse effects to niclosamide
3. Renal impairment
4. Hepatic impairment
5. Pregnancy or a desire to become pregnant
6. Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-12-03 (Estimated); Study Completion 2021-12-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Cure of the patient | 7 days
  To assess the percentage of cure of the patient and evaluated by normalization of clinical evaluation, laboratory investigations, and imaging.
Time to recovery | 7 days
  - to study the time to recovery ( stay days in hospital)

SECONDARY OUTCOMES:
The percentage of Progressive patients | 7 days
  - T assess percentage of progressive patients to more advanced disease
Rate of mortality | 7 days
  - To evaluate mortality rate among NCS add on group compared to controls
Side effects | 7 days
  - To demonstrate side effects seen during the trial and will be assessed according clinical evaluation and the appropriate laboratory investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Abdulamir, Professor, Principal Investigator — College of Medicine-Al-Nahrain University; Faiq I. Gorial, Prof, Principal Investigator — College of Medicine-University of Baghdad; Manal K abdulrrazaq, Professor, Study Chair — College of Medicine-University of Baghdad
Locations (1):
- Ahmed S. Abdulamir, Baghdad, Baghdada, Iraq

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Time Frame: 6 months after publication
Access Criteria: Will be given by the principle investgator